CLINICAL TRIAL: NCT05520879
Title: Community-based Management of Acute Malnutrition (CMAM) in Bangladesh: Effectiveness Trial of Locally Developed Ready-to-use Therapeutic Food in the Treatment of Severe Acute Malnutrition in Rohingya Camps in Cox's Bazar
Brief Title: Effectiveness Trial of Locally Developed Ready to Use Therapeutic Food
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: UNICEF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PR-21014
Record Dates: First submitted 2022-05-19; First posted 2022-08-30 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Malnutrition Severe
Keywords: Severe Acute Malnutrition; Local RUTF; Effectiveness Trial; Forcibly Displaced Myanmar Nationals; Bangladesh
MeSH Terms: conditions — Severe Acute Malnutrition

STUDY DESIGN:
Intervention Model Description: Sharnali-1 and Sharnali-2 would be provided among 450 severely acute malnourished children divided into two groups to assess the proportion of children graduating from SAM to non-acute malnutrition status (MUAC ≥ 125 mm or WLZ/WHZ ≥ -2 for two consecutive weeks) by 90 days of intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention study products will be packaged in sachets that cannot be differentiated between the two.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- To provide Sharnali-1 to severe acute malnourished children (Experimental): We will provide Sharnali-1 among 225 severe acute malnourished children to assess the proportion of children graduating from SAM to non-acute malnutrition status (MUAC ≥ 125 mm or WLZ/WHZ ≥ -2 for two consecutive weeks) by 90 days of intervention.
  Interventions: Dietary Supplement: Sharnali 1
- To provide Sharnali-2 to severe acute malnourished children (Experimental): We will provide Sharnali-2 among 225 severely acute malnourished children to assess the proportion of children graduating from SAM to non-acute malnutrition status (MUAC ≥ 125 mm or WLZ/WHZ ≥ -2 for two consecutive weeks) by 90 days of intervention.
  Interventions: Dietary Supplement: Sharnali 2

INTERVENTIONS:
Dietary Supplement: Sharnali 1 — The intervention is food product, made from locally available food ingredients in Bangladesh.
  Sharnali 1 made from rice, lentil, dried skimmed milk, sugar, vegetable oils and micronutrient premix.
  Arms: To provide Sharnali-1 to severe acute malnourished children
Dietary Supplement: Sharnali 2 — Sharnali 2 made from chick peas, dried skimmed milk, sugar, vegetable oils and micronutrient premix.
  Arms: To provide Sharnali-2 to severe acute malnourished children

SUMMARY:
As poor health conditions and malnutrition are major issues confronting the influx of Forcibly Displaced Myanmar Nationals (FDMN), there is an urgent need to prepare the service providers to control the situation and to prevent deaths and disabilities in FDMN children suffering from severe acute malnutrition (SAM). It is therefore imperative to assess the effectiveness of the two local Nutrition Managements (NMs); Sharnali 1 & Sharnali 2 for the treatment of SAM in an emergency in Bangladesh.

If the effectiveness trial shows that the NMs are effective, either one or both varieties can be used for children with SAM in emergency situations. Ultimately a Bangladeshi solution will replace the expensive RUTF that is currently being imported for use in the FDMN camps for management of SAM.

DETAILED DESCRIPTION:
In response to the huge global burden of childhood acute malnutrition, WHO and UNICEF have recommended since 2007 ready-to-use therapeutic food (RUTF) as the treatment for children with severe acute malnutrition (SAM) without complications in the community. Although there is no national program in Bangladesh for management of SAM in the community, the Ministry of Health and Family Welfare (MoHFW) has posited for a therapeutic food to manage childhood malnutrition that is made of locally available food ingredients. With this backdrop, icddr,b developed two types of such food called Nutritional Management (NM) for the management of uncomplicated SAM in the community. These NMs conform to the National Guidelines on Community-based Management of SAM of the Government of Bangladesh as well as WHO and UNICEF specifications. These newly developed therapeutic foods, named as Sharnali-1 and Sharnali-2, are made of locally available food ingredients including rice, lentils, and chickpeas respectively and a recently conducted trial assessing their acceptability among SAM children showed that the local Bangladeshi NMs are as acceptable as the imported RUTF (Annex1: Composition of the locally developed NMs). Same group of researchers also completed a randomized, double-blind efficacy trial among children with SAM in Dhaka and in Kurigram that revealed that the local NMs are as efficacious as the imported RUTF.

Poor health conditions and malnutrition are major issues confronting the influx of about 1000,000 Forcibly Displaced Myanmar Nationals (FDMN; the FDMN people from across the border into Bangladesh). It is unfortunately anticipated that the deadliest form of malnutrition - severe acute malnutrition (SAM) - will greatly exceed the current national prevalence as a result of severe food insecurity, disease, and the existing high levels of malnutrition among those who are crossing the border. There is an urgent need to prepare ourselves to control the situation and to prevent deaths and disabilities in refugee children suffering from SAM. It is therefore imperative to assess the effectiveness of the two local NMs for the treatment of SAM in an emergency situation in Bangladesh, the FDMN situation being one that demands urgent attention. If the effectiveness trial shows that the NMs are effective, either one or both varieties can be used for children with SAM in emergency situations where food insecurity is extreme. Ultimately, a Bangladeshi solution will replace the expensive RUTF that is currently being imported for use in the FDMN FDMN camps. On the other hand, researchers also want to explore their perception, belief and practices if NMs and RUTF in that community is being provided. Unexpectedly, there is no data available on how they perceive about SAM management and how they would response if the above mentioned services are implemented. Therefore, the researchers would like to explore maternal/caregiver perception, knowledge, practices and barriers towards community-based health care management among FDMN population as well.

The Ministry of Health and Family Welfare of Bangladesh has approved conduction of the trial of the local therapeutic foods, Sharnali-1 and Sharnali-2, developed by icddr,b among under-five children in FDMN Forcibly Displaced Myanmar National (FDMN) camps suffering from SAM.

Objectives:

To assess the effectiveness of two local NMs (Sharnali-1 and Sharnali-2) in managing 6-59 months old children suffering from SAM in the community in an emergency setting (for example, the Camps of Forcibly Displaced Myanmar Nationals).

Methods:

An effectiveness trial will be conducted using the Bangladeshi NMs in the FDMN Camps in Teknaf and Ukhiya sub-districts of Cox's Bazar district. The primary outcome variable of the effectiveness trial is to assess the proportion of children graduating from SAM to non-acute malnutrition status (MUAC ≥ 125 mm or WLZ/WHZ ≥ -2 for two consecutive weeks) by 90 days of intervention. The total number of participants enrolled for the effectiveness trial would be 450 children with SAM in two arms.

ELIGIBILITY:
Inclusion Criteria:

* Severe acute malnourished children
* Age 6-59 months
* Either sex
* No medical complication
* MUAC <115 mm and/or WLZ/WHZ <-3.

Exclusion Criteria:

* Children not suffering from severe acute malnutrition
* Children with oedematous malnutrition
* Failed to obtain consent for study participation from parents or legal guardian
* Suffering from any chronic illness(es) etc.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of children graduating from SAM to non-acute malnutrition status | 90 days
  The primary outcome variable is to assess the proportion of children graduating from SAM to non-acute malnutrition status (MUAC ≥ 125 mm or WLZ/WHZ ≥ -2 for two consecutive weeks) by 90 days of intervention

SECONDARY OUTCOMES:
Time (days) required to graduate from SAM to non-acute malnutrition status | 90 days
  Required Time for graduation from SAM to non acute malnutrition measured in days
Rate of weight gain of children (g/kg per day) during 1st 2 weeks, 1st 4 weeks and up to graduation | 90 days
  Children's weight gain measured as g/kg/day
Proportion of children recovered (MUAC ≥ 125 mm or WLZ/WHZ ≥ -2) by different time periods | 90 days
  Proportion of recovery at different time points measured as percentage
Changes in weight | 90 days
  Changes in body weight measured in kg
Changes in Mid Upper Arm Circumference (MUAC) | 90 days
  Changes in Mid Upper Arm Circumference (MUAC) measured in mm or cm
Changes in height | 90 days
  Changes in height measured in cm
Changes in weight-for-height Z score | 90 days
  Changes in weight-for-height Z score measured in points
Changes in weight-for-age Z score | 90 days
  Changes in weight-for-age Z score measured in points
Changes in height-for-age Z score | 90 days
  Changes in height-for-age Z score measured in points
Proportion of children dropped out | 90 days
  Proportion of children dropped out measured in percentage
Proportion of children relapsed (deterioration of weight, appearance of edema or any clinical emergencies) | 90 days
  Proportion of children relapsed (deterioration of weight, appearance of edema or any clinical emergencies) measured in percentage
Proportion of children needed hospital admission after enrolment | 90 days
  Proportion of children needed hospital admission after enrolment measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Md Munirul Islam, PhD, Study Director — Scientist; Nurun Nahar Naila, MPH, Principal Investigator — Assistant Scientist
Locations (2):
- Bangladesh (2):
  - International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Teknāf, Cox's Bazar
  - International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Ukhiya, Cox's Bazar

IPD SHARING:
Plan to Share IPD: No